CLINICAL TRIAL: NCT02793492
Title: OSPREY ILIAC: Occlusive/Stenotic Peripheral Artery REvascularization StudY for Common And/or External ILIAC Artery Using the Misago® RX Self-expanding Peripheral Stent
Brief Title: Misago® RX Self-expanding Peripheral Stent for Common And/or External Iliac Artery
Acronym: OSPREY ILIAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS2015-01
Record Dates: First submitted 2016-05-16; First posted 2016-06-08 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Iliac Artery Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Misago® RX Self-expanding Stent (Experimental): Eligible participants will undergo stent implantation with the Misago® RX Self-expanding Stent
  Interventions: Device: Misago® RX Self-expanding Peripheral Stent

INTERVENTIONS:
Device: Misago® RX Self-expanding Peripheral Stent — the Misago® RX Self-expanding Stent is a bare metal, nitinol stent

SUMMARY:
This is a multi-center, single arm, non-randomized, prospective clinical study using the Misago® RX Self-expanding Peripheral Stent for treatment of de novo, restenotic, and/or occlusive lesion(s) of the common and/or external iliac artery.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥ 18 years old and of legal consent.
2. Is willing to comply with all follow-up evaluations at the specified times.
3. Subject or subject's legal representative has been informed of and understands the nature of the study and provides signed informed consent to participate in the study.
4. Has a Rutherford Clinical Category Score of 2, 3 or 4.
5. Radiographic evidence of ≥ 50% stenosis or restenosis (from PTA or adjunct therapy, not including stents or stent grafts), or occlusion of target lesion(s) in the common iliac artery and/or external iliac artery.

Exclusion Criteria:

1. Has had previous stent or stent-graft implantation in the target lesion(s).
2. Has a contraindication or known untreatable allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs or any other drug used during the study according to the protocol.
3. Has known hypersensitivity to contrast material that cannot be adequately pretreated.
4. Has known hypersensitivity to nickel-titanium (nitinol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from the composite Major Adverse Event rate, defined as periprocedural related death, amputation of the target limb, and clinically driven TLR assessed at 9 months post-procedure. | 9 months post-procedure

SECONDARY OUTCOMES:
Major Adverse Event rate at 30 days, and 12- and 24- months post-procedure defined as a composite of peri-procedural related death, amputation of the target limb, and clinically driven TLR. | 30 days, 12- and 24- months post-procedure
Primary stent patency at 9 months defined by a binary duplex ultrasound peak systolic velocity ratio ≤ 2.4 at the stented target lesion and absence of TLR. | 9 months post-procedure
Technical Success defined by the following conditions: 1) Successful delivery of the stent at the lesion site 2) Stent(s) successfully deployed in lesion with adequate lesion coverage | The outcome is assessed up to 24 hours from time of enrollment through index procedure.
  Technical success will be evaluated from time of enrollment through index procedure
Procedural Success: Attainment of < 30% residual stenosis of the target lesion and no peri-procedural complications. | The outcome is assessed up to 24 hours from time of enrollment through index procedure
  Procedural success will be evaluated from time of enrollment through index procedure. Peri-procedural complications defined as: death, stroke, myocardial infarction (MI), emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel.
Clinical Success: Relief or improvement (without increase of one or more in the score) from baseline symptoms as measured by the Rutherford score for chronic limb ischemia at 30 days as compared to baseline. | 30 days post-procedure
  Clinical success will be evaluated from time of enrollment through index procedure. In addition, evaluation of Rutherford sustained (without increase of one or more in the score) at 9 months post-procedure from 30 days post-procedure for durability of results.
Ankle Brachial Index (ABI) change from baseline | through 9 months post-procedure
Clinically driven Target Vessel Revascularization (TVR) at 30 days and 9, 12- and 24- months post-procedure | 30 days and 9, 12 and 24 months post-procedure
  TVR is defined as any re-intervention or artery bypass surgery involving the target vessel in which the subject has ≥ 50% diameter stenosis with worsening symptoms, or ≥ 70% stenosis without symptoms. The target vessel is defined as the vessel containing the treated lesion (e.g., common and/or external iliac artery).
Clinically driven TLR through 30 days and 9-, 12- and 24-months post-procedure. | 30 days and 9-, 12- and 24-months post-procedure
  Clinically driven TLR is defined as re-intervention of the target lesion in which subject has ≥ 50% stenosis with worsening symptoms, or ≥ 70% stenosis without symptoms
Walking Impairment Questionnaire | change from baseline (pre-procedure) at 30 days and 9 months post procedure
Evaluation of all AEs | pre-discharge through 24 months post-procedure
Evaluation of access site complications including severe bleeding, hematoma, and pseudoaneurysm, occurring prior to hospital discharge. | The event is assessed from time of enrollment through hospital discharge or up to 7 days post procedure, whichever occurs first
Occurrence of device deficiency | through 24 months post-procedure
  A device deficiency has occurred when there is inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling
Device Related Complications | 9 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: John Rundback, MD, Principal Investigator — Holy Name Medical Center
Locations (9):
- United States (9):
  - ClinRe Inc. Advanced Heart and Vein Center, Thornton, Colorado
  - University of Florida Health, Gainesville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Holy Name Medical Center, Teaneck, New Jersey
  - Novant Health, Matthews, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No